CLINICAL TRIAL: NCT01886586
Title: RECALL: Retaining Cognition While Avoiding Late-Life Depression
Brief Title: Retaining Cognition While Avoiding Late-Life Depression
Acronym: RECALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Meryl Butters, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10110050
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; memory impairment; problem-solving therapy; depression prevention; caregiver stress; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Caregiver Burden; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Problem Solving Therapy (Active Comparator): 8-12 sessions of Problem Solving Therapy (both members of dyad)
  Interventions: Behavioral: Problem Solving Therapy
- Problem Solving Therapy + Exercise (Active Comparator): 6-12 sessions of Problem Solving Therapy + Exercise (both members of dyad)
  Interventions: Behavioral: Problem Solving Therapy + Exercise
- Enhanced Usual Care (Active Comparator): Staff will will document and monitor all mental health treatment (e.g., medications that participant may be taking) and psychotherapy (e.g. counseling or social services).
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Problem Solving Therapy — 6-12 sessions of Problem Solving Therapy (both members of dyad)
  Arms: Problem Solving Therapy
Behavioral: Problem Solving Therapy + Exercise — 6-12 sessions of Problem Solving Therapy + Exercise (both members of dyad)
  Arms: Problem Solving Therapy + Exercise
Other: Enhanced Usual Care — Staff will document and monitor all mental health treatment (e.g., medications that participant may be taking) and psychotherapy (e.g. counseling or social services).
  Arms: Enhanced Usual Care

SUMMARY:
This study will adapt Problem Solving Therapy (PST) for individuals with mild cognitive impairment (MCI) as an intervention for preventing major depression (DEP). PST will be modified so as to be provided to both MCI probands as well as their support person. The primary aim is to examine the effectiveness of PST in individuals with MCI and the support person, at preventing DEP over 12 mos. in MCI probands. We also will examine the effect of exercise on preventing depression.

DETAILED DESCRIPTION:
The Recall Study (Retaining Cognition while Avoiding Late-Life Depression) is a study for adults 60 and older who have noticed mild memory changes in themselves or a loved one. Mild memory changes may feel stressful and therefore increase an individual's risk of developing depression. This research project will test whether Problem Solving Therapy (PST) is successful in preventing major depression for those living with mild cognitive impairments. We will also examine the effect of modest exercise on mood. You will participate in 8 to 12 PST sessions over 16 weeks. All treatments are provided at no cost and there is compensation for participation.

ELIGIBILITY:
MCI participant Inclusion Criteria:

1. => age 60
2. Modified Mini Mental State (3MS) => 80
3. MCI diagnosis
4. Adequate physical and sensory function to undergo NP assessment
5. PHQ-9 score 1-9, with at least one of the cardinal symptoms of depression (low mood or anhedonia) endorsed.

MCI participant Exclusion Criteria:

1. Major Depressive Episode or anxiety disorder within the past 1 year
2. Currently taking an anti-depressant
3. History of Bipolar Disorder or Schizophrenia
4. Drug or alcohol use disorder within 12 months
5. Currently taking anti-anxiety med >4x/week for the past 4 weeks

Support person Inclusion Criteria:

1. => age 18
2. Modified Mini Mental State (3MS) => 80
3. Normal Cognitive Function
4. Adequate physical and sensory function to undergo NP assessment
5. PHQ-9 score 1-9, with at least one of the cardinal symptoms of depression (low mood or anhedonia) endorsed.

Support person Exclusion Criteria:

1. Major Depressive Episode or anxiety disorder within the past 1 year
2. Currently taking an anti-depressant
3. History of Bipolar Disorder or Schizophrenia
4. Drug or alcohol use disorder within 12 months
5. Currently taking anti-anxiety med >4x/week for the past 4 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-07; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of depression or anxiety disorders | 15 months
  PHQ9, prime-MD SCID, GAD7

SECONDARY OUTCOMES:
Change in cognitive function measured by RBANS and DKEFS | 15 months
  RBANS, DKEFS, 3MS, PASS, CAMCI, CIRS-G, RAND-12, LLFDI, SPPB, PSQI, NRS, ISEL, PROMIS, Cornell Services Index, P-GIC, ZARIT, DAS

CONTACTS AND LOCATIONS:
Overall Officials: Meryl Butters, MD, Principal Investigator — University of Pittsburgh; Ariel Gildengers, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Late-Life Evaluation and Treatment Center, Pittsburgh, Pennsylvania
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Gildengers AG, Butters MA, Albert SM, Anderson SJ, Dew MA, Erickson K, Garand L, Karp JF, Lockovich MH, Morse J, Reynolds CF 3rd. Design and Implementation of an Intervention Development Study: Retaining Cognition While Avoiding Late-Life Depression (ReCALL). Am J Geriatr Psychiatry. 2016 Jun;24(6):444-54. doi: 10.1016/j.jagp.2015.10.010. Epub 2015 Nov 18. PMID 27066730